CLINICAL TRIAL: NCT00848445
Title: the Use of Atrial Fibrillation Pacing Therapies in Patients With no Previous History of Atrial Fibrillation: Canadian Atrial Fibrillation Evaluation (CAFE) Study -
Brief Title: Atrial Fibrillation: Canadian Atrial Fibrillation Evaluation (CAFE) Study -
Acronym: CAFE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Dr Lawrence Sterns (PI), Victoria Cardiac Arrythmia Trials
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CAFÉ
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- APP and VRR on (Experimental): APP and VRR turned on at 2 week visit
  Interventions: Device: Guidant Pulsar Max II or Insignia Plus DR; Device: Atrial pacing preference turned on or off
- APP and VRR off (Active Comparator): APP and VRR turned off
  Interventions: Device: Guidant Pulsar Max II or Insignia Plus DR; Device: Atrial pacing preference turned on or off

INTERVENTIONS:
Device: Guidant Pulsar Max II or Insignia Plus DR — market approved pacemaker. programmed per protocol
Device: Atrial pacing preference turned on or off — programing changes in the device

SUMMARY:
To evaluate whether atrial fibrillation (AF) therapies in Guidant Pulsar Max II or Insignia Plus DR have an effect on the occurance of AF in patients with no prior history of AF

DETAILED DESCRIPTION:
This multi-centre, randomized, cross-over, prospective study will evaluate the occurrence of AF with AF pacing therapies programmed on (APP and VRR) and with AF therapies programmed off (APP and VRR) in patients with no known prior history of AF (all patients have a pacing indication). The occurrence of AF as well as time to first event and AF burden (frequecy and duration).

ELIGIBILITY:
Inclusion Criteria:

* No prior history of AF or atrial flutter, primary indication of SSS or AV block for dual chamber pacemaker, confidentiality agreement signed and dated before implant, available for follow-up at the study centre where they were enrolled at the protocol defined intervals, willing and capable of participating in all testing associated with the study, on stable regime of arrhythmia management drugs.

Exclusion Criteria:

* Documented history of AF or atrial flutter, clinically significant ventricular arrhythmias, < 18 yrs old, life expectancy < 1 year or expectation of heart transplantation during the study period, likely to or have received a mechanical tricuspid valve during the study, enrolled in other cardiovascular studies, women who are pregnant, inability or refusal to sign Patient Confidentiality Agreement, inability or refusal to complete the follow-up schedule at the study centre in which they were enrolled, exhibit arrhythmias due to reversible cause eg, digitalis toxicity, hypoxia, transient electrolyte imbalance, acute myocardial infarction or electrocution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2002-10 (Actual); Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To compare the occurrence of AF (>350 bpm) during a period when AF pacing therapies are programmed on (APP and VRR) and during when AF therapies are programmed off. | one year

SECONDARY OUTCOMES:
To compare AF burden between patients with AF therapies programmed on (APP and VRR) and patients with AF pacing therapies turned off (APP and VRR). Burden is defined as the product of the number of AF events and duration of events. To compare the time to | one year

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Sterns, MD, Principal Investigator — Victoria Cardiac Arrythmia trials